CLINICAL TRIAL: NCT03321019
Title: Mechanisms of Airway Protection Dysfunction in Parkinson's Disease
Brief Title: Airway Protective Mechanisms in PD (R01)
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201700959-N; 5R01HD091658-05 (NIH)
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Capsaicin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy controls: Men and women between the ages of 45 and 85 years without Parkinson's disease, or any history of neurologic disorder/disease, head or neck cancer, or chronic respiratory illness.
  Interventions: Drug: Capsaicin; Device: Resistive respiratory loads; Other: Event-related evoked potential using electroencephalography (EEG).; Procedure: Fluoroscopic swallow evaluation
- Parkinson's disease: Men and women between the ages of 45 and 85 years with Parkinson's disease, and without any history of neurologic disorder/disease, head or neck cancer, or chronic respiratory illness.
  Interventions: Drug: Capsaicin; Device: Resistive respiratory loads; Other: Event-related evoked potential using electroencephalography (EEG).; Procedure: Fluoroscopic swallow evaluation

INTERVENTIONS:
Drug: Capsaicin — Participants will inhale aerosolized capsaicin with the goal of this inducing cough and an urge-to-cough.
Device: Resistive respiratory loads — Participants will breath through a mouthpiece. Every 3-5 breaths in, a respiratory load will be applied. Participants will be asked to rate the magnitude of the load.
Other: Event-related evoked potential using electroencephalography (EEG). — The study team will use EEG time-locked to a respiratory occlusion to measure the brain's response to respiratory sensation.
  Other Names: ERP; RREP
Procedure: Fluoroscopic swallow evaluation — Participants will swallow various consistencies of barium under fluoroscopy (moving-picture x-ray) in order to assess swallowing safety and efficiency.
  Other Names: Modified barium swallow

SUMMARY:
This study will collect data on various aspects of airway sensation and function, and determine how it relates to the development of swallowing and cough dysfunction in Parkinson's disease. Participants will be followed over a 3-year period, with once-per-year visits to collect the data.

DETAILED DESCRIPTION:
Aspiration pneumonia (APn) occurs at a disproportionately hig rate in patients with Parkinson's disease (PD) versus healthy age-matched older adults. This is of particular public health concern given that aspiration pneumonia infection is a leading cause of death in persons with PD. The development of APn is multifactorial with aspiration of material from disordered swallowing (dysphagia) without proper cough response being the main contributing factor. These findings reflect the fact that both swallowing and cough are sensorimotor behaviors, and thus require appropriate detection and scaling of a sensory stimulus in order to produce an appropriate motor response.

The long-term goal of this research is to advance the management of airway protection deficits in patients with neurodegenerative disease in order to decrease morbidity and mortality due to aspiration related lung infection. The objective here, which is a critical step in pursuit of that goal, is to further specify the sensory mechanisms associated with airway protection disorders in order to advance the clinical management of these patients. In order to accomplish the objective of this application the study team has identified 3 aims: First, determine relationship(s) between airway somatosensation, reflex cough and swallowing function in people with PD, and how these relationships may change with disease progression, over time. Second, determine whether cortical processing of sensory information is associated with deficits in reflex cough sensitivity or swallowing function in people with PD, and third, to determine how the central neural filtering of airway sensory stimuli may relate to the development of airway protective disorders.

The study team will accomplish these aims in 2 experimental studies. First, the study team will test the magnitude of respiratory resistive loads, in people with PD across a range of disease durations, and in a healthy control group. The study team will measure reflex cough, using a cough-inducing irritant (capsaicin), and swallowing function. The study team will perform these tests at 3 time-points, spaced 10-14 months apart, in order to determine the relationships between respiratory sensation, cough sensitivity and effectiveness, and swallowing function, and how they change with advancing disease duration.

Next the study team will perform electroencephalographic recordings time-locked to paired respiratory stimuli to determine cortical processing of airway sensory information. The study team will measure the amplitude and latency of the sensory evoked potential peaks, and compute ratios of peak amplitude between the first and second paired stimulus in order to determine the degree of sensory gating. The realization of the proposed aims and studies is significant because it is a necessary step in our program of research that is expected to lead to earlier, more accurate identification, as well as targeted interventions for airway protection deficits in PD.

Completion of this research is systematically important for our goal of maintaining adequate airway protective function in PD patients; the results are expected to directly impact reductions in health care costs, morbidity, and mortality related to airway protection deficits.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 45 and 85 years
2. Diagnosis of PD, Hoehn and Yahr stages I - IV, by a fellowship trained neurologist arriving at the diagnosis of PD by applying strict UK brain bank criteria (PD participants only)

Exclusion Criteria:

1. Neurological disorders other than PD (i.e., stroke, etc.)
2. Difficulty complying due to neuropsychological dysfunction (i.e., severe depression)
3. Allergy to capsaicin or hot peppers
4. History of head or neck cancer
5. History of smoking in the past 5 years
6. Any neurological disorder including PD (Healthy control group only)

Ages: 45 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study includes both male and female participants. One study group (control group) will be adults between 45 and 85 years of age without Parkinson's disease. The other group will consist of adults between 45 and 85 years of age with Parkinson's disease diagnosed by a movement disorders trained neurologist, according to UK brain bank criteria.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2023-07-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hegland, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Center for Movement Disorders and Neurorestoration, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment began 12/2017 and ended 2/2022. Participants with Parkinson Disease (PD) were recruited from an IRB-approved clinical database of people with PD. Healthy (non-PD) participants were recruited using advertisement fliers and word-of-mouth. All participants were seen in research space at the outpatient Fixel Institute for Neurological Diseases at the University of Florida.
Period: Overall Study
Arm/Group | Healthy Controls | Parkinson's Disease
Started | 19 | 100
Completed | 19 | 72
Not Completed | 0 | 28
Not completed — Withdrawal by Subject | 0 | 6
Not completed — Lost to Follow-up | 0 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Parkinson's Disease | Total
Number analyzed (Participants) | 19 | 100 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 29 | 35
  >=65 years | 13 | 71 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (8.5) | 69.1 (7.3) | 68.8 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 27 | 39
  Male | 7 | 73 | 80
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19 | 100 | 119
Hoehn &Yahr score (PD only) [Median (Full Range); unit: units on a scale] — The Hoehn & Yahr scale is a commonly used system for describing how the symptoms of Parkinson's disease progress. The scale varies from 0: no sign of disease, to stage 5: needing a wheelchair or bedridden unless assisted. Population: Because the Hoehn & Yahr scale score is a disease-specific measure, it was not completed on the healthy control participants.
  units on a scale
    number analyzed (Participants) | 0 | 100 | 100
    (all) |  | 2 [0 to 5] | 2 [0 to 5]
Disease duration (PD only) [Number; unit: participants] — Disease duration is based on years since the diagnosis of Parkinson's disease. The number of participants in each duration range category (1 - 5 years, 6 - 10 years, and 11 or more years) is reported. Population: Disease duration is specific to Parkinson's participants and not reported for healthy control participants, as there is no disease present.
  participants
    1 - 5 years: number analyzed (Participants) | 0 | 100 | 100
    1 - 5 years |  | 49 | 49
    6 - 10 years: number analyzed (Participants) | 0 | 100 | 100
    6 - 10 years |  | 26 | 26
    11 + years: number analyzed (Participants) | 0 | 100 | 100
    11 + years |  | 25 | 25

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Sensitivity
Description: Slope of perception of resistive load and load resistance: Magnitude estimation of respiratory load (6 - no difficulty inhaling - 20 maximum difficulty inhaling) is plotted on the y-axis and respiratory load (0, 5, 10, 25 & 40 cm H2O loads) is plotted on the x-axis. The slope of the resulting regression line is the measure.
Time Frame: 3 years, three time points (assessed at year 1 visit, year 2 visit, and year 3 visit)
Population: The healthy control group had only 1 visit, whereas the PD group had 3 visits. Thus, the 2nd and 3rd rows in the outcome measure table are pertinent only to the PD participants. The numbers analyzed for the PD group in years 2 and 3 are smaller than year 1 due to participant withdrawals or loss to follow up.
Measure: Mean (Standard Deviation); unit: scores on a scale / CmH2O
Arm/Group | Healthy Controls | Parkinson's Disease
Number analyzed (Participants) | 19 | 100
scores on a scale / CmH2O
  Year 1 visit | 0.22 (0.08) | 0.22 (0.07)
  Year 2 visit (PD only): number analyzed (Participants) | 0 | 91
  Year 2 visit (PD only) |  | 0.21 (0.07)
  Year 3 visit (PD only): number analyzed (Participants) | 0 | 72
  Year 3 visit (PD only) |  | 0.22 (0.06)
Statistical Analysis 1: Comparison: Healthy Controls vs Parkinson's Disease; Healthy controls were compared to PD participants across each of the 3 visits. PD participants were compared between visits 1, 2 and 3; Test type: Other; p < .0001, ANOVA — The p value was adjusted for multiple comparisons using Tukey's method; Degree of freedom - 3, 278; F-statistic = 8.59

2. Primary Outcome: Urge to Cough Sensitivity
Description: Urge to cough sensitivity slope: Slope of the line created by plotting the urge to cough (0 indicating none - 10 indicating maximal) on the y-axis and capsaicin concentration (increasing from 0, 25, 50, 100, 200 micromolar) on the x-axis.
Time Frame: 3 years, three time points (assessed at year 1 visit, year 2 visit, and year 3 visit)
Population: For the PD group, the numbers analyzed in years 2 and 3 of the study reflect loss of participants to either withdrawal or loss to follow up.
Measure: Mean (Standard Deviation); unit: scores on a scale / micromolar capsaicin
Arm/Group | Healthy Controls | Parkinson's Disease
Number analyzed (Participants) | 19 | 100
scores on a scale / micromolar capsaicin
  Year 1 | 0.31 (0.08) | 0.22 (0.08)
  Year 2 (PD only): number analyzed (Participants) | 0 | 91
  Year 2 (PD only) |  | 0.21 (0.09)
  Year 3 (PD only): number analyzed (Participants) | 0 | 72
  Year 3 (PD only) |  | 0.20 (0.09)
Statistical Analysis 1: Comparison: Healthy Controls vs Parkinson's Disease; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.72, ANOVA — Tukey's method was used to control for multiple comparisons; Degrees of freedom - 3. 278; F-statistic = .44

3. Primary Outcome: Penetration-aspiration Scale
Description: Rating of airway intrusion of bolus material during swallowing ranging from 1 (best, no airway invasion) to 8 (worst, silent aspiration).
Time Frame: 3 years, three time points (assessed at year 1 visit, year 2 visit, and year 3 visit)
Population: For the PD group, the numbers analyzed in years 2 and 3 of the study reflect loss of participants to either withdrawal or loss to follow up. In some cases fluoroscopy was not available in the year 2 or 3 visit, so some participants were not included due to no data for those visits. Not that on the Penetration-Aspiration scale used, higher numbers are worse, with the full range being 1 (normal swallow) to 8 (silent aspiration).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Healthy Controls | Parkinson's Disease
Number analyzed (Participants) | 19 | 100
score on a scale
  Year 1 | 1 [1 to 8] | 2 [1 to 8]
  Year 2 (PD only): number analyzed (Participants) | 0 | 89
  Year 2 (PD only) |  | 2 [1 to 8]
  Year 3 (PD only): number analyzed (Participants) | 0 | 70
  Year 3 (PD only) |  | 2 [1 to 8]
Statistical Analysis 1: Comparison: Healthy Controls vs Parkinson's Disease; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.02, ANOVA — Dunnett's T3 method was used to account for multiple comparisons; degrees of freedom: 3, 229; F-statistic = 3.048

4. Secondary Outcome: Cough Peak Flow Rate
Description: Highest airflow rate (in liters per second; L/s) during cough
Time Frame: 3 years, three time points (assessed at year 1 visit, year 2 visit, and year 3 visit)
Population: For the PD group, the numbers analyzed in years 2 and 3 of the study reflect loss of participants to either withdrawal or loss to follow up. The measure (L/s) is airflow - higher is better (indicating more airflow out per second), a measure of cough effectiveness.
Measure: Mean (Standard Deviation); unit: Liters of air per second (L/s)
Arm/Group | Healthy Controls | Parkinson's Disease
Number analyzed (Participants) | 19 | 100
Liters of air per second (L/s)
  Year 1 | 3.17 (1.31) | 3.67 (1.31)
  Year 2 (PD only): number analyzed (Participants) | 0 | 91
  Year 2 (PD only) |  | 3.27 (1.2)
  Year 3 (PD only): number analyzed (Participants) | 0 | 72
  Year 3 (PD only) |  | 3.01 (1.18)
Statistical Analysis 1: Comparison: Healthy Controls vs Parkinson's Disease; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.034, ANOVA — The p value was adjusted in the analysis for multiple comparisons using Tukey's method; Degrees of freedom - 3, 231; F-statistic = 2.939

5. Secondary Outcome: Swallowing Timing
Description: Duration from bolus head passing mandible to laryngeal vestibule closure measured in frames. Data are collected at 33 frames per second.
Time Frame: 3 years, three time points (assessed at year 1 visit, year 2 visit, and year 3 visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Frames
Arm/Group | Healthy Controls | Parkinson's Disease
Number analyzed (Participants) | 19 | 100
Frames
  Year 1 | 6.10 (7.24) | 6.70 (10.22)
  Year 2 (PD only): number analyzed (Participants) | 0 | 89
  Year 2 (PD only) |  | 8.85 (6.63)
  Year 3 (PD only): number analyzed (Participants) | 0 | 70
  Year 3 (PD only) |  | 8.14 (5.32)
Statistical Analysis 1: Comparison: Healthy Controls vs Parkinson's Disease; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.022, ANOVA — Tukey's method was used to adjust for multiple comparisons; Degrees of freedom - 3, 274; F-statistic = 1.494

ADVERSE EVENTS:
Time Frame: Adverse even data were collected at year 1 visit, year 2 visit, and year 3 visit for each participant.
Arm/Group | Healthy Controls | Parkinson's Disease
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/100
Other Adverse Events (participants affected / at risk) | 0/19 | 0/100

LIMITATIONS AND CAVEATS:
This study spanned the time of the global COVID pandemic, so many of the participants lost to follow up, and limited ability to recruit, were a direct result of restrictions put in place between March 2020 and March 2021.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT03321019/Prot_SAP_004.pdf
  • Informed Consent Form: ICF2_longitudinal (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT03321019/ICF_005.pdf
  • Informed Consent Form: longitudinal study (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT03321019/ICF_006.pdf